CLINICAL TRIAL: NCT02996565
Title: Pragmatic Trial Comparing Telehealth Care and Optimized Clinic-Based Care for Uncontrolled High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HealthPartners Institute
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
Keywords: Clinic care; Team-based care; Medication Therapy Management (MTM); Telehealth; Cluster-randomized; Home blood pressure monitoring; Pharmacist
MeSH Terms: conditions — Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Practice Clinic-Based Care (Active Comparator): Patients with uncontrolled hypertension who receive primary care in clinics assigned to the Best Practice Clinic-Based Care intervention.
  Interventions: Other: Best Practice Clinic-Based Care
- Telehealth Care (Active Comparator): Patients with uncontrolled hypertension who receive primary care in clinics assigned to the Telehealth Care intervention.
  Interventions: Other: Telehealth Care

INTERVENTIONS:
Other: Best Practice Clinic-Based Care — Relies primarily on the physician-medical assistant dyad and face-to-face visits to promote:
  1. Improved recognition of uncontrolled BP at primary care encounters,
  2. Therapeutic action to address uncontrolled BP at primary care encounters,
  3. Reliable follow-up visits to re-assess uncontrolled BP every 2-4 weeks.
  Arms: Best Practice Clinic-Based Care
Other: Telehealth Care — All elements of Clinic-Based Care are performed, plus a telemonitoring and pharmacist case management program is offered, specifically:
  1. Referral to care by MTM pharmacist or Nurse Practitioner and receiving a home blood pressure telemonitoring device
  2. Systematic home BP telemonitoring with data transmitted into patient medical record
  3. Systematic home-based care by pharmacist or nurse practitioner via telephone and/or secure email
  Arms: Telehealth Care

SUMMARY:
This pragmatic trial will compare two team-based care models for managing hypertension, Best Practice Clinic-based Care and Telehealth Care with pharmacist management, in a large care system in Minnesota. Clinics in the study are randomized to offer one of the two treatment models to participants with uncontrolled hypertension.

The investigators aim to determine a) whether one model is more effective than the other for lowering patient's blood pressure and b) which model patients prefer.

DETAILED DESCRIPTION:
The objectives of the study are:

Aim 1: Compare the effects of two evidence-based strategies on lowering blood pressure and other outcomes important to patients: best-practice clinic-based care and home-based telehealth care.

* Hypothesis 1.1: Compared with patients in clinics assigned to clinic-based care, patients in clinics assigned to telehealth care will have a 5 mm Hg greater change in systolic blood pressure over 12 months of follow-up.
* Hypothesis 1.2: Compared with patients in clinics assigned to clinic-based care, patients in clinics assigned to telehealth care will report: a) fewer treatment side effects; b) better ratings of patient experience of hypertension care; and c) higher self-monitoring rates and confidence in self-care.

Aim 2: Conduct an evaluation of the reach, adoption, implementation, and maintenance of the telehealth care and clinic-based care interventions using a mixed-methods approach supported by the RE-AIM framework and the Consolidated Framework for Implementation Research (CFIR).

ELIGIBILITY:
Inclusion Criteria:

* Hypertension diagnosis code in medical record, twice in last 24 months
* Attends study clinic for primary care visit within study period with uncontrolled blood pressure
* Systolic blood pressure >=150 mm Hg or Diastolic blood pressure >=95 mm Hg at current visit
* Systolic blood pressure >=150 mm Hg or Diastolic blood pressure >=95 mm Hg at most recent previous visit

Exclusion Criteria:

* Pregnancy
* End Stage Kidney Disease
* Patients in hospice care and patients who permanently reside in a nursing home

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3071 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Margolis, MD, Principal Investigator — HealthPartners Institution
Locations (1):
- HealthPartners Institute, Bloomington, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide a de-identified, individual-level dataset to PCORI if requested at the end of the study. The dataset will be made publicly available and will contain no identifying information.

REFERENCES:
- [Derived] Margolis KL, Crain AL, Pawloski PA, Ziegenfuss JY, Trower NK, Bergdall AR, Beran M, Norton CK, Haugen PK, Rehrauer DJ, Green BB, Solberg LI, Sperl-Hillen JM. Blood Pressure Medication Side Effect Symptoms and Patient Treatment Satisfaction and Adherence. J Am Board Fam Med. 2025 Mar-Apr;38(2):312-329. doi: 10.3122/jabfm.2024.240288R1. PMID 40578923
- [Derived] Margolis KL, Bergdall AR, Crain AL, JaKa MM, Anderson JP, Solberg LI, Sperl-Hillen J, Beran M, Green BB, Haugen P, Norton CK, Kodet AJ, Sharma R, Appana D, Trower NK, Pawloski PA, Rehrauer DJ, Simmons ML, McKinney ZJ, Kottke TE, Ziegenfuss JY, Williams RA, O'Connor PJ. Comparing Pharmacist-Led Telehealth Care and Clinic-Based Care for Uncontrolled High Blood Pressure: The Hyperlink 3 Pragmatic Cluster-Randomized Trial. Hypertension. 2022 Dec;79(12):2708-2720. doi: 10.1161/HYPERTENSIONAHA.122.19816. Epub 2022 Oct 25. PMID 36281763
- [Derived] JaKa M, Bergdall A, Beran MS, Solberg L, Green BB, Andersen J, Kodet A, Norman S, Haugen P, Crain L, Trower N, Sharma R, Rehrauer D, Maeztu C, Margolis K. Reach in a pragmatic hypertension trial: A critical RE-AIM component. Contemp Clin Trials. 2022 Oct;121:106896. doi: 10.1016/j.cct.2022.106896. Epub 2022 Aug 24. PMID 36029952
- [Derived] Margolis KL, Crain AL, Green BB, O'Connor PJ, Solberg LI, Beran M, Bergdall AR, Pawloski PA, Ziegenfuss JY, JaKa MM, Appana D, Sharma R, Kodet AJ, Trower NK, Rehrauer DJ, McKinney Z, Norton CK, Haugen P, Anderson JP, Crabtree BF, Norman SK, Sperl-Hillen JM. Comparison of explanatory and pragmatic design choices in a cluster-randomized hypertension trial: effects on enrollment, participant characteristics, and adherence. Trials. 2022 Aug 17;23(1):673. doi: 10.1186/s13063-022-06611-3. PMID 35978336
- [Derived] Solberg LI, Crain AL, Green BB, Ziegenfuss JY, Beran MS, Sperl-Hillen JM, Norton CK, Margolis KL. Experiences and Perceptions of Patients with Uncontrolled Hypertension Who are Dissatisfied with Their Hypertension Care. J Am Board Fam Med. 2021 Nov-Dec;34(6):1115-1122. doi: 10.3122/jabfm.2021.06.210240. PMID 34772767
- [Derived] Margolis KL, Crain AL, Bergdall AR, Beran M, Anderson JP, Solberg LI, O'Connor PJ, Sperl-Hillen JM, Pawloski PA, Ziegenfuss JY, Rehrauer D, Norton C, Haugen P, Green BB, McKinney Z, Kodet A, Appana D, Sharma R, Trower NK, Williams R, Crabtree BF. Design of a pragmatic cluster-randomized trial comparing telehealth care and best practice clinic-based care for uncontrolled high blood pressure. Contemp Clin Trials. 2020 May;92:105939. doi: 10.1016/j.cct.2020.105939. Epub 2020 Jan 22. PMID 31981712

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened and enrolled during primary care encounters at eligible and randomized primary care clinics in a large integrated health system. Patients were enrolled between November 15, 2017 and April 15, 2019.
Pre-assignment Details: Among 57 primary care clinics screened for eligibility, 36 were excluded (16 no MTM; 20 not using automated BP monitor) and 21 were randomized (17 individual clinics plus 4 clinics as 2 co-located pairs).
  Among 69,480 patients screened in primary care encounters, 3,071 met all inclusion criteria and were enrolled in the study and received care according to the clinic-randomized treatment arm.
Units Other Than Participants: Primary Care Clinics
Groups:
- Best Practice Clinic-Based Care: Patients with uncontrolled hypertension who receive primary care in clinics assigned to the Best Practice Clinic-Based Care intervention.
  Best Practice Clinic-Based Care: Relies primarily on the physician-medical assistant dyad and face-to-face visits to promote:
  1. Improved recognition of uncontrolled BP at primary care encounters,
  2. Therapeutic action to address uncontrolled BP at primary care encounters,
  3. Reliable follow-up visits to re-assess uncontrolled BP every 2-4 weeks.
- Telehealth Care: Patients with uncontrolled hypertension who receive primary care in clinics assigned to the Telehealth Care intervention.
  Telehealth Care: All elements of Clinic-Based Care are performed, plus a telemonitoring and pharmacist case management program is offered, specifically:
  1. Referral to care by MTM pharmacist or Nurse Practitioner and receiving a home blood pressure telemonitoring device
  2. Systematic home BP telemonitoring with data transmitted into patient medical record
  3. Systematic home-based care by pharmacist or nurse practitioner via telephone and/or secure email
Period: Overall Study
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Started (Patients) | 1648; 9 Primary Care Clinics | 1423; 10 Primary Care Clinics
Referred to Intended Provider for Hypertension Follow-up (Intended provider: Medical Assistant for BP check (Best Practice) or MTM Pharmacist (Telehealth Care)) | 1480; 9 Primary Care Clinics | 1060; 10 Primary Care Clinics
Attended Follow-up Within 6 Weeks (With Any Provider Type) | 890; 9 Primary Care Clinics | 887; 10 Primary Care Clinics
Attended Follow-up Within 6 Weeks (With Intended Provider) (Intended provider: Medical Assistant for BP check (Best Practice) or MTM Pharmacist (Telehealth Care)) | 532; 9 Primary Care Clinics | 385; 10 Primary Care Clinics
Completed (Met "per protocol" definition for treatment adherence) | 532; 9 Primary Care Clinics | 275; 10 Primary Care Clinics
Not Completed | 1116; 0 Primary Care Clinics | 1148; 0 Primary Care Clinics

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care | Total
Number analyzed (Participants) | 1648 | 1423 | 3071
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (14.2) | 62.4 (14.2) | 60.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 834 | 805 | 1639
  Male | 814 | 618 | 1432
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 14 | 60
  Not Hispanic or Latino | 1585 | 1386 | 2971
  Unknown or Not Reported | 17 | 23 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 15 | 4 | 19
  Asian | 92 | 121 | 213
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 329 | 265 | 594
  White | 1144 | 988 | 2132
  More than one race | 8 | 7 | 15
  Unknown or Not Reported | 59 | 36 | 95
Highest education level [Count of Participants; unit: Participants] — Population: Data available for baseline survey respondents only
  Participants
    number analyzed (Participants) | 908 | 780 | 1688
    High school, GED, or less | 316 | 247 | 563
    Some college or technical school | 315 | 284 | 599
    4-year college degree | 171 | 137 | 308
    >4-year college degree | 106 | 112 | 218
Employment [Count of Participants; unit: Participants] — Population: Data available for baseline survey respondents only
  Participants
    number analyzed (Participants) | 908 | 785 | 1693
    Full-time | 351 | 231 | 582
    Part-time | 71 | 68 | 139
    Retired | 332 | 350 | 682
    Otherwise not working for pay | 154 | 136 | 290
Annual Income [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Data available for baseline survey respondents only
  Participants
    number analyzed (Participants) | 798 | 683 | 1481
    Less than $20,000 | 164 | 143 | 307
    $20,000 to $49,999 | 258 | 185 | 443
    $50,000 to $99,999 | 231 | 238 | 469
    Greater than or equal to $100,000 | 145 | 117 | 262
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 157.4 (15.4) | 158.8 (15.2) | 158.0 (15.3)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 93.1 (13.8) | 90.0 (13.8) | 91.7 (13.9)
Number of anti-hypertensive medication classes [Mean (Standard Deviation); unit: anti-hypertensive medication classes] | 1.7 (1.1) | 1.7 (1.2) | 1.7 (1.1)
Body Mass Index (BMI) greater than or equal to 30 [Count of Participants; unit: Participants] | 987 | 743 | 1730
Diabetes [Count of Participants; unit: Participants] | 407 | 366 | 773
Cardiovascular disease [Count of Participants; unit: Participants] | 247 | 265 | 512

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure Between Baseline and 12 Months (mm Hg)
Description: Change in systolic BP, collected from medical records
Time Frame: Trajectory over 12 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 1648 | 1423
mm Hg | -17.97 [-19.43 to -16.50] | -18.72 [-20.20 to -17.24]
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority; p = 0.45, planned contrast — The threshold for statistical significance was p = 0.05; The planned contrast compares model-predicted change in SBP from index to 365 days in Telehealth Care vs. Best Practice Clinic-Based Care; Mean Difference (Net) = -0.76, 95% CI 2-sided [-2.84 to 1.33] — adjusted for baseline SBP, baseline DBP, baseline age, sex, Asian race

2. Secondary Outcome: Change in Diastolic BP Between Baseline and 12 Months (mm Hg)
Description: change in diastolic BP, collected from medical records
Time Frame: Trajectory over 12 months
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 1648 | 1423
mm Hg | -9.98 [-10.84 to -9.11] | -9.70 [-10.58 to -8.83]
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — Random coefficients model predicted all EHR-documented DBPs from treatment group, days elapsed from index to each DBP (time) and treatment group by time with random clinic and patient intercepts; p = 0.64, planned contrast — The threshold for statistical significance was p<0.05; The planned contrast compares the model-predicted change in DBP from index to 365 days in Telehealth care vs. index to 365 days in clinic based care; Mean Difference (Net) = 0.28, 95% CI 2-sided [-0.95 to 1.51] — adjusted for baseline SBP, baseline DBP, baseline age, sex, Asian race

3. Secondary Outcome: Number of Participants Who Reporting Monitoring BP at Least 2 Times Per Week at Six Months Follow-up
Description: Patient report of monitoring BP at least 2 times per week
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 673 | 603
Participants | 189 | 265
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — Random coefficients model predicted baseline and 6 month patient-reported outcome from treatment group, time point and treatment group by time with random clinic intercept and patient scale parameter; p < 0.001, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The interaction RR compares the likelihood pf reporting high satisfaction at 6 months relative to baseline in Telehealth care vs. clinic based care; Risk Ratio (RR) = 1.53, 95% CI 2-sided [1.27 to 1.85] — adjusted for baseline DBP, baseline age, sex

4. Secondary Outcome: Number of Participants Who Report High Level of Satisfaction With Hypertension Care at Six Months.
Description: Patient rating of 9-10 vs. 0-8 on a scale of 0 (low satisfaction) to 10 (high satisfaction). Developed from a scale used by Green, et al (2008).
  Citation: Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D,Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008;299:2857-2867. doi:10.1001/jama.299.24.2857
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 678 | 610
Participants | 205 | 241
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.03, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 3, analysis 1]; Risk Ratio (RR) = 1.25, 95% CI 2-sided [1.02 to 1.52] — adjusted for baseline DBP, baseline age, sex

5. Secondary Outcome: Number of Participants Who Are Current Smokers at Twelve Months
Description: Current smoker at 12 months
Time Frame: Baseline to 12 months
Population: The numbers of participants analyzed represent the number of participants with smoking status available in the EHR
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 302 | 218
Participants | 273 | 199
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — Random coefficients model predicted the likelihood that smoking was current 12 months by treatment group with random clinic intercept; p = 0.73, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The risk ratio compares the likelihood of current smoking at 12 months in Telehealth care vs. clinic based care; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.95 to 1.07] — unadjusted

6. Secondary Outcome: Number of Participants Reporting Cough as a Side Effect of Antihypertensive Medications at Six Months
Description: Patient report that side effect is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 656 | 593
Participants | 202 | 212
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.08, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The interaction RR compares the likelihood of reporting the side effect was a problem at 6m relative to baseline in Telehealth vs. clinic based care; Risk Ratio (RR) = 1.17, 95% CI 2-sided [.98 to 1.4] — adjusted for baseline DBP, baseline age, sex

7. Secondary Outcome: Number of Participants Reporting Dizziness as a Side Effect of Antihypertensive Medication at Six Months
Description: Patient report that side effect is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 656 | 593
Participants | 247 | 232
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.18, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 6, analysis 1]; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.95 to 1.29] — adjusted for baseline DBP, baseline age, sex

8. Secondary Outcome: Number of Participants Reporting Frequent Urination as a Side Effect of Antihypertensive Medication at Six Months
Description: Patient report that side effect is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 656 | 593
Participants | 331 | 293
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.77, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 6, analysis 1]; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.87 to 1.11] — adjusted for baseline DBP, baseline age, sex

9. Secondary Outcome: Number of Participants Reporting Leg/Foot Swelling as a Side Effect of Antihypertensive Medication at Six Months
Description: Patient report that side effect is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 656 | 593
Participants | 247 | 208
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.32, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 6, analysis 1]; Risk Ratio (RR) = 0.93, 95% CI 2-sided [0.80 to 1.08] — adjusted for baseline DBP, baseline age, sex

10. Secondary Outcome: Number of Participants Reporting Sexual Symptoms as a Side Effect of Antihypertensive Medication at Six Months
Description: Patient report that side effect is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 656 | 593
Participants | 174 | 132
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.62, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 6, analysis 1]; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.76 to 1.19] — adjusted for baseline DBP, baseline age, sex

11. Secondary Outcome: Number of Participants Reporting Tiredness as a Side Effect of Antihypertensive Medication at Six Months
Description: Patient report that side effect is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 656 | 593
Participants | 437 | 376
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.87, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 6, analysis 1]; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.91 to 1.08] — adjusted for baseline DBP, baseline age, sex

12. Secondary Outcome: Number of Participants Who Report Decreasing Salt as Helpful for BP Self-management at Six Months
Description: Patient report that activity is helpful for BP self-management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 538 | 471
Participants | 274 | 242
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.51, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The interaction RR compares the likelihood of reporting the activity is helpful at 6m relative to baseline in Telehealth care vs. clinic based care; Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.82 to 1.11] — adjusted for baseline DBP, baseline age, sex

13. Secondary Outcome: Number of Participants Who Report Limiting Alcohol as Helpful for BP Self-management at Six Months
Description: Patient report that activity is helpful for BP self-management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 339 | 289
Participants | 147 | 138
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.41, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 12, analysis 1]; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.87 to 1.37] — adjusted for baseline DBP, baseline age, sex

14. Secondary Outcome: Number of Participants Who Report Physical Activity as Helpful for BP Self-management at Six Months
Description: Patient report that activity is helpful for BP self management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 560 | 506
Participants | 291 | 256
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.18, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The interaction RR compares the likelihood of reporting the activity was helpful at 6m relative to baseline in Telehealth care vs. clinic based care; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.77 to 1.06] — adjusted for baseline DBP, baseline age, sex

15. Secondary Outcome: Number of Participants Who Report Reducing Stress as Helpful for BP Self-management at Six Months
Description: Patient report that activity is helpful for BP self management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 566 | 482
Participants | 278 | 243
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.31, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 12, analysis 1]; Risk Ratio (RR) = 0.92, 95% CI 2-sided [0.78 to 1.09] — adjusted for baseline DBP, baseline age, sex

16. Secondary Outcome: Number of Participants Who Report Watching Weight as Helpful for BP Self-management at Six Months
Description: Patient report that activity is helpful for BP self management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 556 | 488
Participants | 290 | 249
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.56, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 12, analysis 1]; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.89 to 1.22] — adjusted for baseline DBP, baseline age, sex

17. Secondary Outcome: Number of Participants Identifying Clinic Visits as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 632 | 578
Participants | 196 | 149
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.08, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The interaction RR compares the likelihood of reporting the burden was a problem at 6m relative to baseline in Telehealth care vs. clinic based care; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.68 to 1.03] — adjusted for baseline DBP, baseline age, sex

18. Secondary Outcome: Number of Participants Identifying Cost of Care or Medications as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 649 | 588
Participants | 188 | 134
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.32, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 0.9, 95% CI 2-sided [.73 to 1.11] — adjusted for baseline DBP, baseline age, sex

19. Secondary Outcome: Number of Participants Reporting Increasing Physical Activity as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 615 | 552
Participants | 236 | 242
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.09, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 1.14, 95% CI 2-sided [0.98 to 1.33] — adjusted for baseline DBP, baseline age, sex

20. Secondary Outcome: Number of Participants Reporting Lifestyle Changes as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 601 | 529
Participants | 251 | 192
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.77, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.83 to 1.16] — adjusted for baseline DBP, baseline age, sex

21. Secondary Outcome: Number of Participants Reporting Measuring BP as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 587 | 558
Participants | 158 | 164
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.09, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 1.21, 95% CI 2-sided [.97 to 1.5] — adjusted for baseline DBP, baseline age, sex

22. Secondary Outcome: Number of Participants Reporting Phone Visits as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 479 | 481
Participants | 94 | 66
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.02, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 0.64, 95% CI 2-sided [0.45 to 0.92] — adjusted for baseline DBP, baseline age, sex

23. Secondary Outcome: Number of Participants Reporting Scheduling Visits as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 639 | 579
Participants | 186 | 127
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.006, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 0.70, 95% CI 2-sided [.55 to .89] — adjusted for baseline DBP, baseline age, sex

24. Secondary Outcome: Number of Participants Reporting Time Away From Work as BP Care Burden at Six Months
Description: Patient report that burden is a problem
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 590 | 531
Participants | 159 | 92
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.06, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 17, analysis 1]; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.60 to 1.01] — adjusted for baseline DBP, baseline age, sex

25. Secondary Outcome: Number of Participants Reporting High Confidence in Reporting Contacting Care Team at Six Months Confidence in Managing Blood Pressure: Contact Care Team
Description: Patient reported "very" or "extremely" confident in this aspect of BP management.
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 671 | 598
Participants | 481 | 467
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.65, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The interaction RR compares the likelihood of reporting very/extremely confident at 6m relative to baseline in Telehealth care vs. clinic based care; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.94 to 1.10] — adjusted for baseline DBP, baseline age, sex

26. Secondary Outcome: Number of Participants Reporting High Confidence in Keeping BP Below Target at Six Months
Description: Patient reported "very" or "extremely" confident in this aspect of BP management.
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item.
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 670 | 599
Participants | 242 | 252
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.83, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 25, analysis 1]; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.83 to 1.25] — adjusted for baseline DBP, baseline age, sex

27. Secondary Outcome: Number of Participants Reporting High Confidence in Knowing BP Target Numbers at Six Months
Description: Patient reported "very" or "extremely" confident in this aspect of BP management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 662 | 594
Participants | 437 | 465
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.41, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 25, analysis 1]; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.95 to 1.13] — adjusted for baseline DBP, baseline age, sex

28. Secondary Outcome: Number of Participants Reporting High Confidence in Measuring BP at Home at Six Months
Description: Patient reported "very" or "extremely" confident in this aspect of BP management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 652 | 597
Participants | 376 | 412
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.40, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 25, analysis 1]; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.94 to 1.16] — adjusted for baseline DBP, baseline age, sex

29. Secondary Outcome: Number of Participants Reporting High Confidence in Taking BP Medications at Six Months
Description: Patient reported "very" or "extremely" confident in this aspect of BP management
Time Frame: Baseline to 6 months
Population: The numbers of participants analyzed represent the number of survey respondents who answered the specific survey item
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 667 | 595
Participants | 564 | 532
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.74, Mixed Models Analysis — The threshold for statistical significance was p<0.05; [statistical method as in outcome 25, analysis 1]; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.95 to 1.07] — adjusted for baseline DBP, baseline age, sex

30. Secondary Outcome: Number of Participants With Statin Addition at 12 Months
Description: New statin medication current at 12 months
Time Frame: Baseline to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
Number analyzed (Participants) | 1648 | 1423
Participants | 162 | 151
Statistical Analysis 1: Comparison: Best Practice Clinic-Based Care vs Telehealth Care; Test type: Superiority — Random coefficients model predicted the likelihood that a new statin was current at 12 months by treatment group with random clinic intercept; p = 0.71, Mixed Models Analysis — The threshold for statistical significance was p<0.05; The risk ratio compares the likelihood of a new statin medication that is current at 12 months in Telehealth care vs. clinic based care; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.81 to 1.37] — adjusted for baseline SBP , baseline DBP, baseline age, sex, Asian race

ADVERSE EVENTS:
Time Frame: 2 years
Description: AEs were defined by primary diagnosis codes from outpatient, inpatient, or emergency encounters, active problem list entry, or abnormal lab values. SAEs were defined by primary diagnosis codes from inpatient or emergency encounters.
  AEs and SAEs (hypotension, hypokalemia, hyperkalemia, hyponatremia and abnormal eGFR) were only monitored in those without evidence in the EHR of these conditions in the year prior to study enrollment. The entire study population was monitored for mortality.
Arm/Group | Best Practice Clinic-Based Care | Telehealth Care
All-Cause Mortality (participants affected / at risk) | 42/1648 | 43/1423
Serious Adverse Events (participants affected / at risk) | 29/1646 | 34/1422
Other Adverse Events (participants affected / at risk) | 597/1648 | 567/1422
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Best Practice Clinic-Based Care (N=1646) | Telehealth Care (N=1422)
hypotension (Vascular disorders) | 23/1574 | 26/1360
hypokalemia (Metabolism and nutrition disorders) | 2/1510 | 1/1294
hyperkalemia (Metabolism and nutrition disorders) | 1/1588 | 2/1363
hyponatremia (Metabolism and nutrition disorders) | 3/1535 | 6/1262
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Best Practice Clinic-Based Care (N=1648) | Telehealth Care (N=1422)
hypotension (Vascular disorders) | 119/1574 | 118/1360
hypokalemia (Metabolism and nutrition disorders) | 194/1510 | 187/1294
hyperkalemia (Metabolism and nutrition disorders) | 87/1588 | 105/1363
hyponatremia (Metabolism and nutrition disorders) | 172/1535 | 190/1262
abnormal eGFR (Renal and urinary disorders) | 227/1380 | 219/1122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/65/NCT02996565/Prot_SAP_001.pdf